CLINICAL TRIAL: NCT01533064
Title: Response of Psychiatric Outpatients to the Great East Japan Earthquake
Status: Completed | Type: Observational
Sponsor: Ashikaga Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Funayama Michitaka, Department of Neuropsychiatry, Ashikaga Red Cross Hospital, Ashikaga Red Cross Hospital
Other Study IDs: ARCH 8 2012
Record Dates: First submitted 2012-02-11; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Mood Disorders
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Psychiatric Outpatients

SUMMARY:
Objective: Reports have described how hospitalized psychiatric patients respond to disasters; however, few reports have described the response to disaster among psychiatric outpatients, who have relatively mild disease in comparison with hospitalized, severely ill psychiatric patients. Here the investigators have analyzed the response to disaster among this under-studied population.

Method: The Great East Japan Earthquake on March 11, 2011, was a catastrophic disaster. The investigators studied psychiatric change among a population of psychiatric outpatients in Tochigi prefecture, located ~160 km (~100 miles) southeast of the Fukushima nuclear power plant, in an area that suffered moderate damage from the earthquake. A total of 328 psychiatric outpatients were enrolled and were grouped into the diagnostic categories F2 (schizophrenic, schizotypal, and delusional disorders), F3 (affective disorders), and F4 (neurotic, stress-related, and somatoform disorders). All diagnoses were made using International Classification of Diseases (ICD) 10 criteria. Changes in symptoms were measured as a change in psychotropic medication after the disaster.

DETAILED DESCRIPTION:
Patient progress was determined by whether a change in medication was needed. We focused on psychotropic drug use, including the use of neuroleptics, antidepressants, and benzodiazepines, directly after the disaster on March 11, 2011. Changes in other psychotropic drugs that are prescribed less frequently, such as lithium or anticonvulsants, were not considered in this study. Changes in symptoms that did not require a need to change psychotropic medications were not considered as part of a patient's progress. Physicians rated the relationship between each change in psychotropic drug and the disaster as direct, indirect, or not relevant. Only when three physicians rated the relationship as direct did we consider the change in a patient's progress to be due to the earthquake. Worsening or improvement of symptoms was defined as a change in psychotropic medications as a result of the deterioration or improvement, respectively, of symptoms. The data were stratified by disease category and sex and analyzed using chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of Ashikaga Red Cross Hospital before the Great East Japan Earthquake on March 11, 2011 who are classified as F2 (schizophrenic, schizotypal, and delusional disorders), F3 (affective disorders), or F4 (neurotic, stress-related, and somatoform disorders), using International Classification of Diseases (ICD) 10 diagnostic criteria

Exclusion Criteria:

* Outpatients who did not consult with our hospital in the 2 months after the earthquake were excluded.

Ages: 11 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: a total of 328 psychiatric outpatients of Ashikaga Red Cross Hospital
Sampling Method: Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2011-03; Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Patient progress determined by whether a change in medication was needed. | 2 months after the disaster

CONTACTS AND LOCATIONS:
Overall Officials: Michitaka Funayama, M.D., Principal Investigator — Ashikaga Red Cross Hospital
Locations (1):
- Ashikaga Red Cross Hospital, Ashikaga, Tochigi, Japan